CLINICAL TRIAL: NCT06780904
Title: Comparing the Efficacy of Dry Needling Combined with Passive Stretching and Muscle Energy Technique on Upper Trapezius Myofascial Trigger Points Associated with Neck Pain
Brief Title: Comparing Efficacy of Dry Needling Combined with Passive Stretching and Muscle Energy Technique on Myofascial Trigger Points
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Peradeniya (Other)
Responsible Party: Principal Investigator, M.D.M.T.D.Dissanayake, Physiotherapist, University of Peradeniya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPTAHS
Record Dates: First submitted 2024-12-31; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Neck Pain
Keywords: myofascial trigger points; passive stretching; dry needling; Muscle Energy Technique (MET); Randomized clinical trial; Upper trapezius
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded (Participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group 1 (Active Comparator): Dry needling + Passive stretching
  Interventions: Procedure: Dry Needling
- Treatment group 2 (Other): Dry needling + Muscle Energy technique
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Dry Needling — Treatment protocol:
  1. Dry needling: Prone position, identify trigger points in upper trapezius, use Hong technique with 50mm/0.25 gauge needle, eliciting local twitch response.
  2. Passive stretching: Supine position, cervical spine stretched just short of restriction, hold for 30s with 20s rest, repeat 3 times.
  3. Muscle Energy Technique: Supine position, identify restriction barrier, move spine away from barrier, instruct patient to isometrically contract opposing movement (25% strength), hold for 7-10s, then stretch towards new barrier for 30s, repeat 3 times.
  Other Names: Passive Stretching, Muscle energy Technique

SUMMARY:
The goal of this clinical trial is to assess and compare the efficacy of dry needling (minimally invasive treatment by using a tiny needle) combined with two types of stretching techniques in patients with neck pain for more than 3 months. The main questions it aims to answer are:

Which combination of treatment will 1.give faster relief of pain? 2.improve neck range of motion? and 3.improve disability level of a person with neck pain.

Participants who are interested will be selected according to eligibility criteria. Participants will be divided into two groups. Initially researcher will assess and interview the participants. Two groups will receive two different combinations of interventions. Pre and post measurements will be obtained and then treatment efficacy will be assessed.

DETAILED DESCRIPTION:
46 participants who are interested in this study will be recruited by using convenient sampling method and according to the inclusion and exclusion criteria. Participants then will be divided into two groups by using opaque sealed envelop method.

Initially participants will be interviewed an outcome measures will be taken. As outcome measures Pain will be assessed by using Visual Analogue Scale (VAS), Disability level will be assessed by using Neck Disability Index(NDI), and Neck Range of Motion will be measured by using Universal Goniometer. Participants will receive interventions, two times per week for two weeks. Soon after the last intervention, same outcome measures will be taken again.

Statistical Package for Social Science (SPSS) version 27 (IBM, USA) for Windows will be used for data analysis. The data will be examined using exploratory statistics, and the distributions will be inspected for violations of normality using graphical methods and the Shapiro-Wilk test. Descriptive statistics of the demographic variables and test measurements will be calculated. Based on the satisfaction or violation of normal distribution assumptions, pain intensity (VAS), neck ROMs, pain intensity, and Neck Disability Index (NDI) will be analyzed using parametric or non-parametric tests. Baseline data for pain intensity, neck ROMs and NDI and pain intensity will be compared between the two intervention groups using paired t-test or Wilcoxon signed-rank test. The difference-in changes in each outcome relative to the baseline between intervention groups will be compared using paired t-test or Wilcoxon signed-rank test

ELIGIBILITY:
Inclusion Criteria:

* Presence of neck pain for at least 3 months or more
* Presence of trigger points in the upper trapezius muscle, either unilaterally or bilaterally
* Age between 18 and 60 years

Exclusion Criteria:

* Having an ongoing infection or fever
* Presence of shoulder pathology, such as tendinopathy, impingement syndrome, capsulitis, or bursitis
* History of direct trauma to the shoulder or neck
* Immunosuppressed individuals (e.g., those with cancer)
* Pregnant or recently delivered
* Diagnosis of fibromyalgia
* History of previous neck or shoulder surgery
* Previous local steroid injection or acupuncture
* Any abnormality that restricts cervical range of motion (e.g., degenerative changes, cervical spine spondylolisthesis, disc protrusion, extrusion, or sequestration observed in MRI)
* Uncontrolled diabetes mellitus
* Needle phobia
* Metal allergies
* Cervical instability
* Presence of local skin lesions or infections
* Significant cognitive impairment or uncooperative behavior
* Participants who have previously undergone any form of physiotherapy intervention for the treatment of neck pain or related conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Neck pain | 2 weeks
  Visual Analog Scale (VAS) 0: Represents the minimum value, such as "no pain" or "no discomfort." 100: Represents the maximum value, such as "worst pain imaginable" or "extreme discomfort.

SECONDARY OUTCOMES:
Neck Range of Motion | 2 weeks
  Neck flexion, Extension, Side flexion to affected side, Side flexion to unaffected side, Rotation to affected side and Rotation to unaffected side
Neck disability level | 2 weeks
  Neck Disability Index Structure: Contains 10 items, each scored on a 0-5 scale Scoring: Total score ranges from 0 to 50, Higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Kandy, Kandy, Central Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No